CLINICAL TRIAL: NCT07393555
Title: A Randomized Phase II Study of Sacituzumab Govitecan Alone, Ivonescimab Alone, or Sacituzumab Govitecan and Ivonescimab in Participants With Previously-Treated Actionable Genomic Alteration Positive Stage IV or Recurrent Non-Small Cell Lung Cancer (Lung-MAP Sub-Study)
Brief Title: Treatment for Advanced Non-small Cell Lung Cancer With Actionable Genomic Alterations After Targeted Treatment and Chemotherapy (An Expanded Lung-MAP Treatment Trial)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S1900N; NCI-2026-00250 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1900N (Other: SWOG); S1900N (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Lung Non-Small Cell Carcinoma; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Specimen Handling; Magnetic Resonance Spectroscopy; sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1 (ivonescimab, sacituzumab govitecan) (Experimental): Patients receive ivonescimab IV over 1-2 hours on day 1 of each cycle and sacituzumab govitecan IV over 1-3 hours on day 1 and 8 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Ivonescimab; Procedure: Magnetic Resonance Imaging; Biological: Sacituzumab Govitecan
- Arm 2 (sacituzumab govitecan) (Experimental): Patients receive sacituzumab govitecan IV over 1-3 hours on day 1 and 8 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Biological: Sacituzumab Govitecan
- Arm 3 (ivonescimab) (Experimental): Patients receive ivonescimab IV over 1-2 hours on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Ivonescimab; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Biological: Ivonescimab — Given IV
  Other Names: AK 112; AK-112; AK112; Anti-PD-1/Anti-VEGF Bispecific Antibody AK112; Anti-PD-1/VEGF Bispecific Antibody AK112; PD-1/VEGF Bispecific Antibody AK112; SMT 112; SMT-112; SMT112
  Arms: Arm 1 (ivonescimab, sacituzumab govitecan); Arm 3 (ivonescimab)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Sacituzumab Govitecan — Given IV
  Other Names: hRS7-SN38 Antibody Drug Conjugate; IMMU 132; IMMU-132; IMMU132; RS7 SN38; RS7-SN38; RS7SN38; Sacituzumab Govitecan-hziy; Trodelvy
  Arms: Arm 1 (ivonescimab, sacituzumab govitecan); Arm 2 (sacituzumab govitecan)

SUMMARY:
This phase II Expanded Lung-MAP treatment trial compares how well sacituzumab govitecan alone, ivonescimab alone, or sacituzumab govitecan in combination with ivonescimab works in treating patients with non-small cell lung cancer (NSCLC) that has come back after a period of improvement (recurrent) or is stage IV and has a change in at least 1 of these genes: ALK, EGFR, HER2 (ERBB2), MET, NTRK, RET, and ROS1. This type of gene change is called an actionable genomic alteration (AGA), which means certain treatments can target the change to fight the cancer. Sacituzumab govitecan is a monoclonal antibody, called sacituzumab, linked to a toxic drug called SN-38. Sacituzumab govitecan is a form of targeted therapy because it attaches to specific molecules (receptors) on the surface of tumor cells, known as TROP2 receptors, and delivers SN-38 to kill them. Ivonescimab is a bispecific antibody that can bind to two different antigens at the same time. It binds to programmed cell death protein 1 (PD1), a protein found on the surface of T cells (a type of white blood cell) and vascular endothelial growth factor (VEGF), a protein found on the surface of tumor cells. Ivonescimab may strengthen the immune system and interfere with the ability of tumor cells to grow and spread. Giving a combination of sacituzumab govitecan and ivonescimab work better than either drug alone, and sacituzumab govitecan alone, ivonescimab alone, or sacituzumab govitecan and ivonescimab together may work better than standard treatments at shrinking NSCLC with an AGA.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare progression-free survival (PFS) between participants randomized to the combination of sacituzumab govitecan plus ivonescimab (SG-I) and sacituzumab govitecan (SG) alone. (Comparison between arms) II. To compare progression-free survival (PFS) between participants randomized to SG-I and ivonescimab (I) alone. (Comparison between arms) III. To evaluate the response (confirmed and unconfirmed, complete and partial) rate of SG against historical response rates. (Single Arm evaluation) IV. To evaluate the response (confirmed and unconfirmed, complete and partial) rate of I against historical response rates. (Single Arm evaluation) V. To evaluate the response (confirmed and unconfirmed, complete and partial) rate of SG-I against historical response rates. (Single Arm evaluation)

SECONDARY OBJECTIVES:

I. To evaluate the rate of dose-limiting toxicities among participants treated with SG-I in the safety run-in analysis population.

II. To compare response rates between ivonescimab with or without sacituzumab govitecan.

III. To compare response rates of sacituzumab govitecan with or without ivonescimab.

IV. To compare overall survival between the SG-I and SG arms. V. To compare overall survival between the SG-I and I arms. VI. To summarize disease control rates within each treatment arm. VII. To summarize the duration of response (DoR) among responders within each treatment arm.

VIII. To evaluate the central nervous system (CNS) progression-free survival per local investigator assessment in participants with baseline CNS metastasis within each treatment arm.

VIII. To evaluate the frequency and severity of toxicities within each treatment arm.

IX. To evaluate if clinical outcomes (response, progression-free survival [PFS], overall survival [OS]) within each treatment arm differs between the subgroup of participants with EGFR mutations to those without EGFR mutations.

X. To evaluate if clinical outcomes (response, PFS, OS) within each treatment arm differs between the subgroup of participants by the presence or absence of PD-L1 expression (< 1% vs 1% or greater).

TRANSLATIONAL MEDICINE OBJECTIVES:

I. To perform comprehensive next-generation sequencing of circulating tumor deoxyribonucleic acid (DNA) (ctDNA) at baseline in all participants to assess its clinical utility in comparison to tumor tissue biomarker profiles.

II. To process and bank cell free DNA (cfDNA) at cycle 3 day 1 and progression for future development of a proposal to evaluate comprehensive next-generation sequencing of circulating tumor DNA (ctDNA).

III. To establish a tissue/blood repository to pursue future studies.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM 1: Patients receive ivonescimab intravenously (IV) over 1-2 hours on day 1 of each cycle and sacituzumab govitecan IV over 1-3 hours on day 1 and 8 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) or magnetic resonance imaging (MRI) and blood sample collection throughout the study.

ARM 2: Patients receive sacituzumab govitecan IV over 1-3 hours on day 1 and 8 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI and blood sample collection throughout the study.

ARM 3: Patients receive ivonescimab IV over 1-2 hours on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI and blood sample collection throughout the study.

After completion of study treatment, patients without disease progression are followed every 12 weeks or more often as clinically indicated until progression, then every 6 months for 2 years and then at end of 3 years from date of randomization. Patients with disease progression are followed every 6 months for 2 years and then at end of 3 years from date of randomization.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have been assigned to S1900N by the Southwest Oncology Group (SWOG) Statistics and Data Management Center (SDMC). Assignment to S1900N is determined by submission of documentation of NSCLC harboring an actionable genomic alteration (AGA) in the LUNGMAP protocol. AGA is defined in this protocol as an activating driver alteration with an approved targeted therapy for lung cancer in one of the following genes: ALK, EGFR, HER2 (ERBB2), MET, NTRK, RET, and ROS1.
* Participants must have measurable disease documented by CT or MRI. The CT from a combined positron emission tomography (PET)/CT may be used to document only non-measurable disease unless it is of diagnostic quality. Measurable disease must be assessed within 28 days prior to randomization. Pleural effusions, ascites and laboratory parameters are not acceptable as the only evidence of disease. Non-measurable disease must be assessed within 42 days prior to randomization. All disease must be assessed and documented on the Baseline Tumor Assessment Form. Participants whose only measurable disease is within a previous radiation therapy port must demonstrate clearly progressive disease (in the opinion of the treating investigator) prior to randomization.
* Participants must have a CT or MRI scan of the brain to evaluate for CNS disease within 42 days prior to randomization.
* Participants with spinal cord compression or brain metastases must not have residual neurological dysfunction, unless no further recovery is expected, and the participant has been stable on weaning doses of corticosteroids (≤ 10 mg daily prednisone or equivalent) prior to randomization. Participants with spinal cord compression or brain metastases that require local treatment must have received local treatment to these metastases and remained clinically controlled and asymptomatic for at least 7 days following stereotactic radiation and/or 14 days following whole brain radiation, and prior to randomization.
* Participants must not have leptomeningeal disease that requires CNS-specific treatment prior to randomization and must not be planning to receive the CNS-specific treatment while on study.
* Participants must have progressed (in the opinion of the treating physician) during or following the most recent line of systemic therapy.
* Participants must have previously received an appropriate targeted therapy for the lung cancer AGA (ALK, EGFR, HER2 (ERBB2), MET, NTRK, RET, and ROS1).
* Participants must have previously received platinum-based chemotherapy for stage IV or recurrent disease.
* Participants must have received no more than (<=) 3 lines of prior cytotoxic therapy (including chemotherapy, antibody-drug conjugates) for NSCLC.
* Participants must not have received prior TROP2-targeted antibody-drug conjugate or a systemic therapy containing sacituzumab govitecan/SN-38.
* Participants must not have received prior anti-PD-1 or anti-PD-L1 antibody therapy.
* Participants must not have received any systemic lung cancer therapy (except orally administered drugs) within 21 days prior to randomization. Orally administered lung cancer therapies must not have been administered within 10 days prior to randomization.
* Participants must have completed any prior radiation therapy within 7 days prior to randomization.
* Participants must have recovered (≤ Grade 1) from any side effects of prior therapy (except for alopecia) prior to randomization.
* Participants must not be planning to receive any concurrent systemic therapy (e.g. chemotherapy, immunotherapy, targeted therapy etc) for lung cancer treatment while receiving treatment on this study.
* Participants' most recent Zubrod performance status must be 0-1 and be documented within 28 days prior to randomization.
* Participants must have a complete medical history and physical exam within 28 days prior to randomization.
* Absolute neutrophil count ≥ 1.5 x 10^3/uL (within 28 days prior to randomization)
* Hemoglobin >= 10.0 g/dL (within 28 days prior to randomization)
* Platelets ≥ 100 x 10^3/uL (within 28 days prior to randomization)
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) unless history of Gilbert's disease (within 28 days prior to randomization). Participants with history of Gilbert's disease must have total bilirubin ≤ 5 x institutional ULN.
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × institutional ULN (within 28 days prior to randomization). Participants with history of liver metastasis must have AST and ALT ≤ 5 x ULN
* Participants must have calculated creatinine clearance ≥ 50 mL/min using the following Cockcroft-Gault Formula. This specimen must have been drawn and processed within 28 days prior to randomization.
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, must have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants must be class 2B or better.
* Participants must not have experienced an arterial or venous thrombotic event or hemoptysis within 28 days prior to randomization.
* Participants must not be planning to receive warfarin (or other coumadin derivatives) while receiving treatment on this study.
* Participants must not have a prior or concurrent malignancy whose natural history or treatment (in the opinion of the treating physician) has the potential to interfere with the safety or efficacy assessment of the investigational regimen.
* Participants must not be pregnant or nursing (nursing includes breast milk fed to an infant by any means, including from the breast, milk expressed by hand, or pumped). Individuals who are of reproductive potential must have agreed to use an effective contraceptive method with details provided as a part of the consent process. A person who has had menses at any time in the preceding 12 consecutive months or who has semen likely to contain sperm is considered to be of "reproductive potential." In addition to routine contraceptive methods, "effective contraception" also includes refraining from sexual activity that might result in pregnancy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) including hysterectomy, bilateral oophorectomy, bilateral tubal ligation/occlusion, and vasectomy with testing showing no sperm in the semen.
* Participants with known human immunodeficiency virus (HIV)-infection must be on effective anti-retroviral therapy and have undetectable viral load test on the most recent test results obtained within 6 months prior to randomization.
* Participants with evidence of chronic hepatitis B virus (HBV) infection must have undetectable HBV viral load while on suppressive therapy on the most recent test results obtained within 6 months prior to randomization.
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. Participants currently being treated for HCV infection must have undetectable HCV viral load test on the most recent test results obtained within 6 months prior to randomization.
* Participants must agree to have blood specimens submitted for circulating tumor DNA (ctDNA)
* Participants must be offered the opportunity to participate in specimen banking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2026-08-07 (Estimated); Primary Completion 2028-11-30 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) (Comparison between arms) | From date of randomization to date of first documentation of progression, symptomatic deterioration, or death due to any cause, assessed up to 3 years
  Will compare between participants randomized to the combination of sacituzumab govitecan plus ivonescimab (SG-I) and sacituzumab govitecan (SG) alone. The comparison of PFS will be done using a 1-sided 10% level log-rank test stratified by randomization stratification factors. Binary proportions along with 90% confidence intervals will be estimated for response to be consistent with 1-sided 5% level testing. With 35 participants per arm, binary proportions can be estimated to within 11% with 90% confidence. The distribution PFS will be estimated using the method of Kaplan-Meier. Comparisons of event time distributions between arms will be summarized by hazard ratios and 80% confidence intervals (consistent with 1-sided 10% level testing) from a Cox Proportional hazards model including the stratification factors.
PFS (Comparison between arms) | From date of randomization to date of first documentation of progression, symptomatic deterioration, or death due to any cause, assessed up to 3 years
  Will between participants randomized to SG-I and ivonescimab (I) alone. The comparison of PFS will be done using a 1-sided 10% level log-rank test stratified by randomization stratification factors. Binary proportions along with 90% confidence intervals will be estimated for response to be consistent with 1-sided 5% level testing. With 35 participants per arm, binary proportions can be estimated to within 11% with 90% confidence. The distribution PFS will be estimated using the method of Kaplan-Meier. Comparisons of event time distributions between arms will be summarized by hazard ratios and 80% confidence intervals (consistent with 1-sided 10% level testing) from a Cox Proportional hazards model including the stratification factors.
Response rate of SG against historical response rates (Single arm evaluation) | Up to 3 years
  Within each treatment arm, the objective is to evaluate if response rates show activity beyond standard of care, which generally would be single agent chemotherapy or docetaxel combined with ramucirumab. With 35 eligible and evaluable participants per arm, the evaluation has 90% exact power to rule out a 10% response rate using a 1-sided 5% level test (the exact level is 5.1% based on design assumptions), if the true response rate were at least 29%. The observation of at least 7 participants with a response (a 20% response rate) would be considered evidence to rule out a 10% response rate.
Response rate of I against historical response rates (Single arm evaluation) | Up to 3 years
  Within each treatment arm, the objective is to evaluate if response rates show activity beyond standard of care, which generally would be single agent chemotherapy or docetaxel combined with ramucirumab. With 35 eligible and evaluable participants per arm, the evaluation has 90% exact power to rule out a 10% response rate using a 1-sided 5% level test (the exact level is 5.1% based on design assumptions), if the true response rate were at least 29%. The observation of at least 7 participants with a response (a 20% response rate) would be considered evidence to rule out a 10% response rate.
Response rate of SG-I against historical response rates (Single arm evaluation) | Up to 3 years
  Within each treatment arm, the objective is to evaluate if response rates show activity beyond standard of care, which generally would be single agent chemotherapy or docetaxel combined with ramucirumab. With 35 eligible and evaluable participants per arm, the evaluation has 90% exact power to rule out a 10% response rate using a 1-sided 5% level test (the exact level is 5.1% based on design assumptions), if the true response rate were at least 29%. The observation of at least 7 participants with a response (a 20% response rate) would be considered evidence to rule out a 10% response rate.

SECONDARY OUTCOMES:
Rate of dose-limiting toxicities among participants treated with SG-I in the safety run-in analysis population | During the first cycle of treatment (21 days)
  Defined as treatment-related Grade 3 or higher non hematologic toxicity, treatment-related Grade 4 or higher hematologic toxicity, or any Grade of treatment-related toxicity that leads to drug discontinuation. Toxicities will be graded based on Common Terminology Criteria for Adverse Events (CTCAE).
Response rates | Up to 3 years
  Will compare response rates between I with or without SG.
Response rates | Up to 3 years
  Will compare response rates between SG with or without I.
Overall survival (OS) | From date of randomization to date of death due to any cause, assessed up to 3 years
  Will compare between the SG-I and SG arms. The distribution of OS will be estimated using the method of Kaplan-Meier. Comparisons of event time distributions between arms will be summarized by hazard ratios and 80% confidence intervals (consistent with 1-sided 10% level testing) from a Cox Proportional hazards model including the stratification factors.
OS | From date of randomization to date of death due to any cause, assessed up to 3 years
  Will compare between the SG-I and I arms. The distribution of OS will be estimated using the method of Kaplan-Meier. Comparisons of event time distributions between arms will be summarized by hazard ratios and 80% confidence intervals (consistent with 1-sided 10% level testing) from a Cox Proportional hazards model including the stratification factors.
Duration of response (DoR) | From date of first documentation of response to date of first documentation of progression, symptomatic deterioration, or death due to any cause among participants who achieve a response, assessed up to 3 years
  The distribution of DoR will be estimated using the method of Kaplan-Meier.
Central nervous system (CNS) PFS | From date of randomization to date of first documentation of progression, symptomatic deterioration, or death due to any cause, assessed up to 3 years
  CNS progression is defined as the development of new CNS metastasis or progression of CNS disease requiring either local CNS therapy or a change in systemic cancer therapy. The distribution of CNS PFS will be estimated using the method of Kaplan-Meier. Comparisons of event time distributions between arms will be summarized by hazard ratios and 80% confidence intervals (consistent with 1-sided 10% level testing) from a Cox Proportional hazards model including the stratification factors.
Frequency and severity of toxicities | During the first cycle of treatment (21 days)
  Toxicities will be graded based on Common Terminology Criteria for Adverse Events (CTCAE). Toxicities will be summarized as proportions by item and worst grade reported, among those possible, probably, or likely related to treatment and also grouped overall and as hematologic and non-hematologic toxicities. Any toxicity, with at least 10% true prevalence has a 97% chance of being observed.
Clinical outcomes by EGFR subgroups | Up to 3 years
  Subgroup analyses will be done using a Cox proportional hazards model for time-to-event outcomes and logistic regression for binary endpoints.
Clinical outcomes by PD-L1 expression subgroups | Up to 3 years
  Subgroup analyses (PD-L1 expression [< 1% vs 1% or greater]) will be done using a Cox proportional hazards model for time-to-event outcomes and logistic regression for binary endpoints.

CONTACTS AND LOCATIONS:
Overall Officials: Susan C Scott, Principal Investigator — SWOG Cancer Research Network